CLINICAL TRIAL: NCT01465906
Title: Efficacy and Safety of Tulobuterol Patch Combined With Tiotropium Bromide for Relieving Dyspnea Symptom of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Chunxue Bai, Director of Respiratory Department , Shanghai Zhongshan Hospita, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG1015TLT
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tulobuterol; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tulobuterol combined with tiotropium bromide (Experimental)
  Interventions: Drug: tulobuterol; Drug: tiotropium bromide
- Tiotropium bromide (Active Comparator)
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: tulobuterol — patch, 2mg, qN, 3 months
  Arms: tulobuterol combined with tiotropium bromide
Drug: Tiotropium Bromide — 18ug, inhale, qD, 3 months
  Arms: Tiotropium bromide
Drug: tiotropium bromide — 18ug, inhale, qD, 3 months
  Arms: tulobuterol combined with tiotropium bromide

SUMMARY:
Phrase: IV

Indication: dyspnea symptom of chronic obstructive pulmonary disease (COPD)

Objective: to evaluate efficacy and safety of tulobuterol patch combined with Tiotropium bromide for relieving dyspnea symptom of COPD

Design: a multi-centre randomized parallel blank control study

Case number: test group 80, control group 80, totally 160

Site number:7

Study period: 2010.9 - 2011.8

ELIGIBILITY:
Inclusion Criteria:

* people aging from 40 to 80 with self ability of judgment
* out-patients diagnosed as stable COPD according to "diagnosing and treatment guideline of COPD (2007 edition)" by Respiratory Department of Chinese Medical Association
* PFT value at screen phase meet the standard as follows: FEV1/FVC < 70% and FEV1% among 30%-80% 15 mins after inhalation of 400ug Ventolin (i.e., moderate and severe COPD patients ).
* people who can use Tiotropium Bromide powder inhalation device
* people who join the study voluntarily and sign ICF (Informed Consent Form)

Exclusion Criteria:

* people who have other acute or chronic respiratory diseases which may cause impairment of pulmonary function such as asthma
* AECOPD （acute exacerbation of COPD）
* people who got respiratory failure 1 month before the study
* people who received oral corticoid treatment 1 month before the study
* people who undergo oxygen therapy at home because of respiratory failure
* people who are allergic to β2 receptor agonist such as tulobuterol
* patients with Skin diseases such as atopic dermatitis, who are not appropriate to use transdermal patch
* patients of hyperthyroidism, hypertension, heart disease and severe arrhythmia, diabetes mellitus, who are not appropriate to useβ2 receptor agonist
* patients who have undergone pulmonary lobectomy or have tumor
* active tuberculosis patients
* people who got acute respiratory tract infection in a month or during screening phase
* allergic rhinitis patients
* glaucoma patients
* people who have diseases which may cause dysuria such as prostatic hypertrophy or bladder neck occlusion
* gestation, lactation and child-bearing age women who don't agree to take contraceptive measures during the study
* people with abnormal live or kidney function, people with nervous system diseases, malignant tumor, neutropenia or other progressive basic diseases.
* People who are mental retardation, mentally ill, deaf-mute or uncooperative, who cannot correctly describe their disease or do corresponding respiratory questionnaire.
* People who are allergic to atropine and its derivatives (including tiotropium bromide and ipratropium bromide), lactose or any inhalant components.
* people who have taken part in other medical clinical trial
* other conditions that investigators think not appropriate for the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
PFT values (pulmonary function test, see description below) | 3 months
  IC (inspiratory capacity) 、PEF (peak expiratory flow)、FVC (forced vital capacity)、FEV1 (forced expiratory volume in the first second)、%FEV1 (forced expiratory volume in the first second as predicted)、RV (residual volume)、TLC (total lung capacity)、RV/TLC% (residual volume/total lung capacity as percentage), etc.
MRC （Medical Research Council） grade | 3 months

SECONDARY OUTCOMES:
SGRQ （St. George's questionnaire） score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, doctor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China